CLINICAL TRIAL: NCT03848000
Title: Randomised Controlled Feasibility Study to Examine the Efficacy of a Combined Group-based Exercise and Educational Programme on Alcohol Consumption, Mental Health and Physical Health Among Alcohol-Dependent Adults
Brief Title: Examination of Whether an Exercise Programme Reduces Alcohol Consumption Among Alcohol-Dependent Adults
Acronym: AOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other); University of Hertfordshire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Active over Alcohol study
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Abuse or Dependence; Alcohol Use Disorder
Keywords: Alcohol abuse; Exercise; Alcohol consumption; Depression; Anxiety
MeSH Terms: conditions — Alcoholism; Motor Activity; Alcohol Drinking; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Programme and NHS Standard Care (Experimental): Exercise and NHS standard care.
  Interventions: Other: Exercise Programme; Behavioral: NHS Standard Care
- NHS Standard Care only (Active Comparator): Alcohol addiction counselling.
  Interventions: Behavioral: NHS Standard Care

INTERVENTIONS:
Other: Exercise Programme — Two sessions per week for 12 consecutive weeks. 30 minute education talks covering topics regarding the physical and mental health benefits of exercise and behaviour change. The following 30-60 minute exercise sessions will utilise pad-boxing, football, body-weight training and circuit training.
  Arms: Exercise Programme and NHS Standard Care
Behavioral: NHS Standard Care — Weekly one-to-one cognitive-behavioral counselling alcohol addiction support session lasting 1 hour. Drug therapy will be offered if indicated in line with standard therapy.

SUMMARY:
This study is composed of two phases. Phase 1 will determine baseline demographic characteristics of participants, currently drinking harmful amounts of alcohol, who would be interested in an alternative treatment option to reduce alcohol consumption. Once baseline data is collected, participants will then be informed that the intervention is an exercise programme and those interested will be offered participation in Phase 2: a two-arm randomised controlled study. If eligible, participants will be randomly assigned to either: 1) a 12 week combined exercise programme and NHS standard care group, or 2) 12 weeks of NHS (National Health Service) standard care only group.

The aims are to study the feasibility of conducting a randomised controlled trial in this cohort and to determine the effectiveness of the exercise programme to reduce alcohol consumption, improve physical and mental health among people drinking harmful amounts of alcohol, compared to standard NHS care. Assessment visits, measuring alcohol consumption, mental health and physical health, will be conducted at baseline, and at Weeks 13, 24, 36 and 48 since commencement of the intervention period. Focus groups will take place during the 2nd and 12th week of the exercise programme where qualitative feedback on the exercise programme will be collected.

DETAILED DESCRIPTION:
Alcohol-dependent patients often experience depression, anxiety and stress, and it is thought that these may be important factors associated with increased alcohol consumption. Regular moderate/high-intensity exercise has been repeatedly reported to reduce depression, anxiety and stress, with regular exercise also shown to be effective in achieving a pleasurable state, improving coping mechanisms and increasing self-confidence among substance-dependent patients. Additionally, exercise-based therapy may be perceived by alcohol-dependent patients as a less stigmatising therapy option than traditional medication and counselling treatments.

While a small number of studies suggest that regular exercise is effective in improving fitness levels among alcohol-dependent adults, there is a lack of consensus regarding the efficacy of regular exercise to reduce alcohol consumption. Of a recent systematic review, 3 of the 5 studies reported that regular exercise reduced alcohol consumption and craving of alcohol. However, while a recent meta-analysis didn't find evidence of exercise significantly reducing alcohol consumption, the three small studies that were assessed all found that exercise training induced some reductions in alcohol consumption; suggesting that regular exercise may be effective in reducing alcohol consumption.

This study is composed of two phases. Phase 1 will determine the characteristics of participants currently drinking harmful amounts of alcohol who would be interested in being offered a new, alternative treatment to reduce alcohol consumption. During their NHS standard care (Phase 1; Visit 1), potential participants will be asked by either a member of the study team, or by the standard care team, if they "would you be willing to consider taking part in a study to look at new ways of treating people addicted to alcohol?'. While no specific details of the intervention will be provided at this time, participants who are interested will be given the participant information sheet (Phase 1) which will include further details of the study. A member of the study team will contact potential participants and, if they are happy to take part, another visit (Phase 1; Visit 2) will be arranged for patients to complete the demographic questionnaires. Visit 2 will take place at one of the study sites and written informed consent will be taken before the patient completes the study questionnaires which will determine characteristics including age, gender, ethnicity, marital status, educational background, employment status, smoking status, number of previous attempts to reduce alcohol consumption, family history of addiction, other drug intake, alcohol consumption (7 Day Drinking Diary), dependence of alcohol consumption (Alcohol Use Disorders Identification Test (AUDIT) questionnaire), severity of alcohol dependence (SADQ), alcohol craving (Penn Alcohol Craving Scale), impact of alcohol consumption on daily life (Alcohol Problems Questionnaire), depression (Patient Health Questionnaire (PHQ-9)), anxiety (Generalised Anxiety Disorder (GAD-7) questionnaire) and current physical activity levels (short-form International Physical Activity Questionnaire (IPAQ)).

Participants who complete Phase 1 of the study will be invited to participate in Phase 2 of the study on the same day (i.e. at the end of Visit 2 of Phase 1 of the study). Interested participants will be provided with full information regarding the nature of the randomised controlled trial - i.e. that this is an exercise-based intervention study - and will be given a separate participant information sheet (Phase 2). A member of the study team will contact potential participants and, if they are happy to participate, the screening visit will be arranged. Participants who decline enrolment into the exercise-based randomized controlled trial will be asked if they are willing to take part in a short telephone interview to enquire about reasons for not wanting to partake in the study. Both participants who agree, and do not agree, to take part in the short telephone interview will be offered NHS standard care. The telephone interviews will be audio-recorded, with participants consent, and transcribed verbatim. This will allow us to identify the characteristics of participants who are interested in exercise. Baseline demographics and characteristics of participants offered the intervention, who consent to provision of data, will be recorded and compared to the demographics of those who decline to participate in the intervention.

Participants who agree to participate in Phase 2 of the study will undergo screening for eligibility. Written informed consent for Phase 2 of the study will be undertaken with a 2nd informed consent form. This visit will be conducted by a member of the study team at one of the NHS hospital sites and current medications and medical history will be recorded, as well as the Physical Activity Readiness Questionnaire (PARQ), to provide a screening measure of physical readiness for exercise. Only if the participant meets the inclusion/exclusion criteria will they be allowed to continue into the study. Participants who do not meet the inclusion/exclusion criteria will be informed that they are not eligible and will be offered NHS standard care. At the end of the screening visit, an accelerometer (Actigraph) will be provided to participants who will be asked to wear it for seven consecutive days in order to measure baseline physical activity levels.

Participants will return the accelerometer (from the screening visit) during the baseline testing visit and will complete the Alcohol Self-Efficacy Scale, Perceived Stress Scale and Short Form (SF-36) questionnaire, before having all physical health measurements (resting heart rate, resting blood pressure, stature, body mass, waist circumference, cardiorespiratory fitness) recorded. A venous blood sample will be collected to measure full blood count and liver enzyme biomarkers, while a finger-prick capillary blood sample will be collected to measure phosphatidylethanol (PEth); a marker of alcohol consumption.

Once the baseline testing visit is completed, participants will be randomly assigned to one of two groups: 1) a 12 week combined exercise (moderate/high-intensity) programme and NHS standard care group (n=48), or 2) 12 weeks of NHS standard care only group (n=48).

The exercise programme will take place in a local sports centre facility in East London, and will be delivered by qualified exercise coaches linked to West Ham United Football Club. Participants will be required to complete two sessions each week for 12 consecutive weeks, in addition to receiving NHS standard care consisting of counselling and support. Each session will begin with a 30 minute education talk (covering topics regarding the physical and mental health benefits of exercise and behaviour change) and will be followed by a 30-60 minute exercise session. Each exercise session will begin with a standard low-intensity 10 minute warm-up/stretch and end with a low-intensity 5 minute cool-down. The main body of the exercise session will utilise a combination of different exercise modalities, including pad-boxing, football and circuit training. The duration of exercise sessions will be gradually increased as follows: Weeks 1-2: 30 minutes; Weeks 3-4: 40 minutes; Weeks 5-6: 50 minutes; Weeks 7-12: 60 minutes. Recruitment of participants will be split into three separate intakes and each exercise group will consist of approximately 15 patients. Participants in the exercise programme will be invited to participate in focus groups on the 3rd session (week 2) and 24th session (week 12) of the exercise programme. The two focus groups will each last approximately 1 hour each and will be conducted by a member of the study team who is fully trained and experienced in undertaking focus group discussions. During the week 2 focus group, the topics for discussion will be the participant's knowledge and beliefs regarding exercise, their barriers to being physically active, their attitude and motivation to being physically active, their expectations of the exercise programme, and what challenges they foresee during the programme. During the week 12 focus group, the topics for discussion will be the participant's experience of the programme, the potential benefits of the programme and what impact it has had on their alcohol consumption, physical health and quality of life. The focus groups will be audio-recorded, with patients consent, and fully transcribed verbatim, anonymized and coded. A thematic analysis will be undertaken to identify recurring and salient themes that are conceptually and inherently significant.

Participants who are randomised to the NHS standard care only group will not receive the exercise programme but will be provided with NHS standard care at one of the NHS study sites. Participants will be provided with the name of their alcohol key worker and will receive a weekly one-to-one counselling alcohol addiction session lasting 1 hour where support and behavioural interventions will be offered, in line with current NHS practice. Drug therapy will be offered if indicated in line with standard therapy.

At the completion of the 12 week intervention period, participants in both the combined exercise programme and NHS standard care group, and the NHS standard care only group will complete 4 follow-up testing visits: at Week 13, Week 24, Week 36 and Week 48 after commencement of the study. These follow-up visits will coincide with the participants routine, clinically-necessary hospital visits. All follow-up visits will be conducted by a member of the study team at one of the NHS hospital sites. At the start of each of the follow-up visits, a member of the study team will verify that the participant is still happy to continue with their participation in the study. Participants will complete the alcohol consumption, physical health, mental health and physical activity questionnaires (the same as the baseline testing visit) at each follow-up testing visit. The finger-prick capillary blood sample, collected to measure phosphatidylethanol (PEth); a marker of alcohol consumption, will only be collected at the Week 24 follow-up visit. At the end of the Week 13 and Week 48 visits, the participant will be given an accelerometer and asked to wear it for seven consecutive days in order to measure physical activity levels over the next week. A visit window of 2 weeks will be set for the Week 13 follow-up testing visit while a visit window of 4 weeks will be set for the Week 24, Week 36 and Week 48 follow-up testing visits to allow for missed or rescheduled appointments.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years old
* AUDIT score of ≥ 8
* In the opinion of the referring physician, is capable of performing moderate/high-intensity exercise
* Agrees to their GP being informed of their participation
* Able and willing to provide written informed consent and complete the study questionnaires

Exclusion Criteria:

* Absolute contraindications to exercise testing and training as defined by the American College of Sports Medicine.
* Have anorexia, bipolar disorder or severe (unstable) psychosis disorder which may preclude active participation.
* In the opinion of the referring physician, is physically incapable or likely to be incapable of undertaking an exercise programme.
* Pregnant or planning pregnancy within the first 3 months after randomisation.
* Currently participating in >90 minutes/week of structured moderate-intensity exercise, such as jogging, cycling or swimming (not including walking).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in absolute total weekly alcohol consumption from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in absolute total weekly alcohol consumption will be assessed by changes in self-reported units of alcohol consumed per week (via a 7 day self-reported drinking diary)
Change in absolute total weekly alcohol consumption from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in absolute total weekly alcohol consumption will be assessed by changes in self-reported units of alcohol consumed per week (via a 7 day self-reported drinking diary)
Change in absolute total weekly alcohol consumption from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in absolute total weekly alcohol consumption will be assessed by changes in self-reported units of alcohol consumed per week (via a 7 day self-reported drinking diary)
Change in absolute total weekly alcohol consumption from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in absolute total weekly alcohol consumption will be assessed by changes in self-reported units of alcohol consumed per week (via a 7 day self-reported drinking diary)

SECONDARY OUTCOMES:
Change in number of drinking days per week from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in the number of drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of drinking days per week from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in the number of drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of drinking days per week from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in the number of drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of drinking days per week from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in the number of drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of heavy drinking days per week from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in the number of heavy drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of heavy drinking days per week from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in the number of heavy drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of heavy drinking days per week from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in the number of heavy drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of heavy drinking days per week from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in the number of heavy drinking days per week will be quantified from a 7 day self-reported drinking diary
Change in number of alcohol free days per week from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in the number of alcohol free days per week will be quantified from a 7 day self-reported drinking diary
Change in number of alcohol free days per week from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in the number of alcohol free days per week will be quantified from a 7 day self-reported drinking diary
Change in number of alcohol free days per week from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in the number of alcohol free days per week will be quantified from a 7 day self-reported drinking diary
Change in number of alcohol free days per week from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in the number of alcohol free days per week will be quantified from a 7 day self-reported drinking diary
Change in Alcohol Use Disorders Identification Test (AUDIT) score from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in Alcohol Use Disorders Identification Test (AUDIT) score will be determined by the completion of a 10-item AUDIT questionnaire
Change in Alcohol Use Disorders Identification Test (AUDIT) score from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in Alcohol Use Disorders Identification Test (AUDIT) score will be determined by the completion of a 10-item AUDIT questionnaire
Change in Alcohol Use Disorders Identification Test (AUDIT) score from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in Alcohol Use Disorders Identification Test (AUDIT) score will be determined by the completion of a 10-item AUDIT questionnaire
Change in Alcohol Use Disorders Identification Test (AUDIT) score from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in Alcohol Use Disorders Identification Test (AUDIT) score will be determined by the completion of a 10-item AUDIT questionnaire
Change in Severity of Alcohol Dependence Questionnaire (SADQ) score from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in the Severity of Alcohol Dependence Questionnaire (SADQ) score will be determined by the completion of the 20-item SADQ questionnaire
Change in Severity of Alcohol Dependence Questionnaire (SADQ) score from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in the Severity of Alcohol Dependence Questionnaire (SADQ) score will be determined by the completion of the 20-item SADQ questionnaire
Change in Severity of Alcohol Dependence Questionnaire (SADQ) score from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in the Severity of Alcohol Dependence Questionnaire (SADQ) score will be determined by the completion of the 20-item SADQ questionnaire
Change in Severity of Alcohol Dependence Questionnaire (SADQ) score from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in the Severity of Alcohol Dependence Questionnaire (SADQ) score will be determined by the completion of the 20-item SADQ questionnaire
Change in alcohol cravings from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in alcohol cravings will be quantified by the completion of the 5-item Penn Alcohol Craving Scale questionnaire
Change in alcohol cravings from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in alcohol cravings will be quantified by the completion of the 5-item Penn Alcohol Craving Scale questionnaire
Change in alcohol cravings from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in alcohol cravings will be quantified by the completion of the 5-item Penn Alcohol Craving Scale questionnaire
Change in alcohol cravings from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in alcohol cravings will be quantified by the completion of the 5-item Penn Alcohol Craving Scale questionnaire
Change in abstinence self-efficacy from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in alcohol abstinence self-efficacy will be determined by the completion of the 40-item Alcohol Abstinence Self-Efficacy Scale questionnaire
Change in abstinence self-efficacy from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in alcohol abstinence self-efficacy will be determined by the completion of the 40-item Alcohol Abstinence Self-Efficacy Scale questionnaire
Change in abstinence self-efficacy from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in alcohol abstinence self-efficacy will be determined by the completion of the 40-item Alcohol Abstinence Self-Efficacy Scale questionnaire
Change in abstinence self-efficacy from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in alcohol abstinence self-efficacy will be determined by the completion of the 40-item Alcohol Abstinence Self-Efficacy Scale questionnaire
Change in alcohol problems from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in social problems caused by alcohol consumption will be determined by the completion of the 49-item Alcohol Problems questionnaire
Change in alcohol problems from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in social problems caused by alcohol consumption will be determined by the completion of the 49-item Alcohol Problems questionnaire
Change in alcohol problems from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in social problems caused by alcohol consumption will be determined by the completion of the 49-item Alcohol Problems questionnaire
Change in alcohol problems from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in social problems caused by alcohol consumption will be determined by the completion of the 49-item Alcohol Problems questionnaire
Change in blood phosphatidylethanol (PEth) from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in blood phosphatidylethanol (collected via finger-prick capillary blood test)
Change in blood gamma glutamyl transferase from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in the liver enzyme biomarker gamma glutamyl transferase (collected during venous blood collection)
Change in blood gamma glutamyl transferase from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in the liver enzyme biomarker gamma glutamyl transferase (collected during venous blood collection)
Change in blood gamma glutamyl transferase from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in the liver enzyme biomarker gamma glutamyl transferase (collected during venous blood collection)
Change in blood gamma glutamyl transferase from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in the liver enzyme biomarker gamma glutamyl transferase (collected during venous blood collection)
Change in blood alanine aminotransferase from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in the liver enzyme biomarker alanine aminotransferase (collected during venous blood collection)
Change in blood alanine aminotransferase from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in the liver enzyme biomarker alanine aminotransferase (collected during venous blood collection)
Change in blood alanine aminotransferase from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in the liver enzyme biomarker alanine aminotransferase (collected during venous blood collection)
Change in blood alanine aminotransferase from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in the liver enzyme biomarker alanine aminotransferase (collected during venous blood collection)
Change in blood aspartate aminotransferase from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in the liver enzyme biomarker aspartate aminotransferase (collected during venous blood collection)
Change in blood aspartate aminotransferase from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in the liver enzyme biomarker aspartate aminotransferase (collected during venous blood collection)
Change in blood aspartate aminotransferase from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in the liver enzyme biomarker aspartate aminotransferase (collected during venous blood collection)
Change in blood aspartate aminotransferase from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in the liver enzyme biomarker aspartate aminotransferase (collected during venous blood collection)
Change in anxiety from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in anxiety scores derived from the 7-item Generalised Anxiety Disorder (GAD-7) Questionnaire
Change in anxiety from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in anxiety scores derived from the 7-item Generalised Anxiety Disorder (GAD-7) Questionnaire
Change in anxiety from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in anxiety scores derived from the 7-item Generalised Anxiety Disorder (GAD-7) Questionnaire
Change in anxiety from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in anxiety scores derived from the 7-item Generalised Anxiety Disorder (GAD-7) Questionnaire
Change in depression from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in depression scores derived from the 9-item Patient Health Questionnaire (PHQ-9)
Change in depression from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in depression scores derived from the 9-item Patient Health Questionnaire (PHQ-9)
Change in depression from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in depression scores derived from the 9-item Patient Health Questionnaire (PHQ-9)
Change in depression from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in depression scores derived from the 9-item Patient Health Questionnaire (PHQ-9)
Change in stress from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in stress scores derived from the 10-item Perceived Stress Scale questionnaire
Change in stress from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in stress scores derived from the 10-item Perceived Stress Scale questionnaire
Change in stress from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in stress scores derived from the 10-item Perceived Stress Scale questionnaire
Change in stress from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in stress scores derived from the 10-item Perceived Stress Scale questionnaire
Change in body weight from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in body weight
Change in body weight from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in body weight
Change in body weight from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in body weight
Change in body weight from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in body weight
Change in cardiorespiratory fitness from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in cardiorespiratory fitness (Chester Step Test)
Change in cardiorespiratory fitness from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in cardiorespiratory fitness (Chester Step Test)
Change in cardiorespiratory fitness from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in cardiorespiratory fitness (Chester Step Test)
Change in cardiorespiratory fitness from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in cardiorespiratory fitness (Chester Step Test)
Change in waist circumference from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in waist circumference
Change in waist circumference from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in waist circumference
Change in waist circumference from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in waist circumference
Change in waist circumference from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in waist circumference
Change in resting systolic and diastolic blood pressure from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in resting systolic and diastolic blood pressure
Change in resting systolic and diastolic blood pressure from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in resting systolic and diastolic blood pressure
Change in resting systolic and diastolic blood pressure from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in resting systolic and diastolic blood pressure
Change in resting systolic and diastolic blood pressure from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in resting systolic and diastolic blood pressure
Change in resting heart rate from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in resting heart rate
Change in resting heart rate from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in resting heart rate
Change in resting heart rate from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in resting heart rate
Change in resting heart rate from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in resting heart rate
Change in objective low-intensity physical activity levels from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in low-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective moderate-intensity physical activity levels from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in moderate-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective high-intensity physical activity levels from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in high-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective very high-intensity physical activity levels from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in very high-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective total physical activity expenditure from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in total physical activity expenditure (kcal/day), as derived from an Actigraph accelerometer
Change in objective sedentary time from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in sedentary time (minutes/day), as derived from an Actigraph accelerometer
Change in objective low-intensity physical activity levels from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in low-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective moderate-intensity physical activity levels from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in moderate-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective high-intensity physical activity levels from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in high-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective very high-intensity physical activity levels from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in very high-intensity physical activity (minutes/day), as derived from an Actigraph accelerometer
Change in objective total physical activity expenditure from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in total physical activity expenditure (kcal/day), as derived from an Actigraph accelerometer
Change in objective sedentary time from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in sedentary time (minutes/day), as derived from an Actigraph accelerometer
Change in subjective physical activity levels from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  Change in vigorous-intensity and moderate-intensity physical activity levels, as determined by the International Physical Activity Questionnaire (IPAQ)
Change in subjective physical activity levels from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  Change in vigorous-intensity and moderate-intensity physical activity levels, as determined by the International Physical Activity Questionnaire (IPAQ)
Change in subjective physical activity levels from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  Change in vigorous-intensity and moderate-intensity physical activity levels, as determined by the International Physical Activity Questionnaire (IPAQ)
Change in subjective physical activity levels from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  Change in vigorous-intensity and moderate-intensity physical activity levels, as determined by the International Physical Activity Questionnaire (IPAQ)
Change in Quality of Life score from baseline, at 13 weeks follow-up | Baseline visit and Week 13 follow-up visit
  The change in quality of life score will be determined by the completion of the 36-item Short Form (SF-36) Questionnaire
Change in Quality of Life score from baseline, at 24 weeks follow-up | Baseline visit and Week 24 follow-up visit
  The change in quality of life score will be determined by the completion of the 36-item Short Form (SF-36) Questionnaire
Change in Quality of Life score from baseline, at 36 weeks follow-up | Baseline visit and Week 36 follow-up visit
  The change in quality of life score will be determined by the completion of the 36-item Short Form (SF-36) Questionnaire
Change in Quality of Life score from baseline, at 48 weeks follow-up | Baseline visit and Week 48 follow-up visit
  The change in quality of life score will be determined by the completion of the 36-item Short Form (SF-36) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Graham R Foster, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No